CLINICAL TRIAL: NCT00193648
Title: Novel Therapies for Resistant FSGS
Brief Title: Pilot Studies of Novel Therapies to Treat Resistant Focal Segmental Glomerulosclerosis (FSGS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: University of North Carolina (Other); The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK70341
Record Dates: First submitted 2005-09-10; First posted 2005-09-19 (Estimated); Last update posted 2007-10-22 (Estimated); Status verified 2007-10

CONDITIONS: Focal Glomerulosclerosis
Keywords: FSGS; Pharmacokinetics; Rosiglitazone; PPAR-gamma agonist; Adalimumab; TNF-alpha antagonist; Steroid and immunosuppressive drug resistance; Resistant primary FSGS
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental | interventions — Rosiglitazone; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Avandia (rosiglitazone)
  Interventions: Drug: Rosiglitazone (Avandia)
- 2 (Active Comparator): Humira (adalimumab)
  Interventions: Drug: Adalimumab (Humira)

INTERVENTIONS:
Drug: Rosiglitazone (Avandia) — oral drug administration
  Arms: 1
Drug: Adalimumab (Humira) — Injection of drug biweekly
  Arms: 2

SUMMARY:
The current management of primary FSGS is predicated on the assumption that the disease is caused by an immune-mediated disturbance in glomerular barrier function. Therefore, most treatment protocols have involved immunosuppressive drugs given singly or in combination. However, the efficacy of this type of therapy has been disappointing and the long-term prognosis for renal survival in patients with resistant FSGS is poor. An alternative approach that targets the fibrosis pathway may represent a novel approach to the treatment of resistant FSGS. In this R21, the investigators will test the hypothesis that two novel agents - a tumor necrosis factor-alpha (TNF-α) antagonist and a peroxisome proliferator activator receptor-gamma (PPARγ) agonist - can be administered safely to patients with resistant FSGS. In the R21 feasibility/pilot phase, pharmacokinetic studies will be conducted to assess the impact of proteinuria on the kinetics of the novel drugs in children and adults.

Specific Aim #1: To assess the safety and tolerability of two novel drugs - a TNF-α antagonist and a PPARγ agonist - in patients with resistant FSGS.

Specific Aim #2: To conduct a pharmacokinetic (PK) assessment of the selected agents to enable selection of medication regimens for investigation in a randomized Phase II study.

DETAILED DESCRIPTION:
Description of study visits

Screening Visit: Eligibility Studies

1. History and physical examination
2. Urine protein and creatinine excretion. Proteinuria (Up/c) will be expressed as the protein:creatinine ratio (mg:mg) in a single early morning specimen.
3. Serum creatinine and calculated GFR. The GFR will be calculated using the Schwartz formula for patients below 18 years of age and Cockroft-Gault for those 18 years or older.
4. Serum Na+, K+, HCO3-, Cl-, glucose, BUN, albumin, cholesterol, AST, ALT, alkaline phosphatase, CBC, ANA, CH50, pregnancy test
5. HIV, Hepatitis B and C serology, if not done in the previous 12 months
6. TB skin test, if not done in the previous 12 months
7. Existing renal biopsy tissue will be assessed for all subjects who have not had the diagnosis of FSGS confirmed by an FSGS-CT core pathologist (only in screen failures).

Baseline Visit: Week 0 Visit

1. Serum glucose, albumin, and creatinine concentrations
2. TNF-alpha level
3. Baseline anti-adalimumab antibody (AAA) level in patients assigned to Humira® treatment
4. A urine, plasma, serum and DNA sample will be collected for storage in the NIDDK FONT Biorepositories at Fisher Bioservice and the Rutgers Cell & DNA Repository for patients who consent to this procedure. A request will be made to store any residual renal tissue collected for clinical indications during the FONT trial in the NIDDK Biorepository.
5. PK assessment (see below)

Follow-up Assessment: Week 2, 4, 8, and 12 Visits

1. Interval history, physical examination, assessment of adverse events
2. Urine protein excretion
3. Serum creatinine and calculated GFR, serum Na+, K+, HCO3, Cl-, glucose, BUN, ALT, AST at all visits
4. Serum albumin, cholesterol, ANA, CH50 at 8-week visit, CBC at all visits except 2-week visit
5. Trough serum adalimumab level in patients assigned to receive Humira® at all visits except 2-week visit
6. Serum AAA level at 12-week visit in patients assigned to Humira® treatment
7. Pregnancy test at 12-week visit

Final Assessment: Week 16 Visit

1. Interval history, physical examination, assessment of adverse events
2. Urine protein excretion
3. Serum creatinine and calculated GFR
4. Serum Na+, K+, HCO3, Cl-, glucose, BUN, albumin, cholesterol, AST, ALT, alkaline phosphatase, CBC, ANA, CH50, and serum TNF-alpha levels
5. Serum AAA level in patients assigned to Humira® treatment
6. Serum, plasma, and urine samples to the NIDDK Biosample Repository at Fisher Bioservice
7. Assessment of patient satisfaction with treatment using TSQM
8. Steady state PK assessment (see below)

The following Table summarizes the laboratory assessment during the R21 study.

Study Medications:

Study medication will be shipped in a single batch sufficient to complete the 4-month treatment period. A supply will be shipped to the participating site for each individual patient that is enrolled. Please complete the Site Registration Form and provide a complete and accurate shipping address for receipt of study medication during the week, Monday though Friday 9 AM - 5 PM. This information will be forwarded to the pharmaceutical companies to enable timely shipment of drug to each site.

Formulation and administration of experimental novel therapies

Adalimumab (Humira®): TNF-α antibody BB-IND #11714:

This medication will be provided by Abbott Laboratories and will be available as a liquid. It will be administered as a subcutaneous injection every other week. The therapeutic dose of adalimumab will be 24 mg/m2 to a maximum of 40 mg/dose every other week for the entire treatment period.

Patients should be instructed to rotate the site of injection. In order to reduce the pain associated with the biweekly adalimumab injections, patients can apply EMLA crème or steroid inhaler spray prior to administration of the medication. After the injection is completed, the patient can take Tylenol as needed or apply ice to the site for symptomatic pain relief.

Patients receiving Humira® will be required to write down dates and times of drug administration and bring the administration log to each study visit. In addition, when a patient is assigned to the Humira® arm, a per protocol dose schedule listing the week and the optimal date of drug administration will be sent with the medication to the site. This sheet can be used to facilitate scheduling of visits and it can be shared with the patient.

Rosiglitazone (Avandia®): PPARgamma agonist IND69,782:

This medication will be provided by Glaxo Smith Kline and will be available as pills. It will be administered orally in two divided daily doses. The therapeutic dose of rosiglitazone will be 3 mg/m2/day administered in two divided doses to a maximum of 4 mg twice a day. The twice daily dosing schedule is based on studies indicating greater antiproteinuric effect of rosiglitazone in type 2 diabetes when administered in this manner.

Pharmacokinetic (PK) Studies

Sampling Scheme:

The blood and urine collection scheme for the PK analysis will be conducted over 48 hours in a GCRC when the patient is scheduled to receive the first dose (single dose PK assessments) of adalimumab or rosiglitazone and after the 8th dose of adalimumab (~steady state of 105 days) or during the 4th month of rosiglitazone therapy for multiple dose PK assessments.

A blood sample, 2.5-4 ml/sample (1-2.5 ml plasma/serum), will be drawn at each time point. For adalimumab, a total of 6 serum samples (4 ml each, 24 ml of blood in total) will be obtained. For rosiglitazone a total of 11 plasma samples (2.5 ml each, 25 ml of blood in total) will be obtained during the 48-hour PK study. The total amount of blood drawn should be < 3 ml/kg over this period.

Urine will be collected at the following intervals: 0-2, 2-12, 12-24, 24-36, and 36-48 hours. The total volume of urine for each time interval should be recorded in mL and an aliquot should be analyzed for protein:creatinine ratio in the local laboratory. The measurements of urinary protein excretion over the 48 hour period will be used to correlate PK parameters of the study medication with concurrent level of proteinuria.

An aliquot of the urine sample collected during each time interval should be saved in the specimen kit for determination of urinary excretion of rosiglitazone. However, because adalimumab cannot be measured in the urine, urinary excretion of the monoclonal antibody will not be performed and an aliquot of urine will NOT be saved in the specimen kit for measurement of Humira®.

If patients must go home after the first day of testing, then they will return to the GCRC on day 2 for repeat blood draws and to return urine collections.

The exact sampling times (hours) for the 48-hour PK studies for each novel therapy, which coincide with the midpoint of the urine collections (see below), are outlined in the following Table:

DRUG 0 0.5 1 2 4 6 8 12 18 30 42 Adalimumab X X X X X X Rosiglitazone* X X X X X X X X X X X

* Serum glucose concentration will be measured at each time point.

Trough serum adalimumab levels should be drawn at 1 week after the first dose of the drug as part of the PK study but not as part of a formal patient visit. In addition to the PK studies, trough serum adalimumab levels will also be drawn prior to the dose at the 2-, 4-, 8-, and 12-week visits.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 2-42 years at onset of proteinuria
2. Aged ≤ 42 years at time of randomization (randomization date before 43rd birthday)
3. Estimated glomerular filtration rate (GFR) ≥ 40 ml/min/1.73 m2 at most recent measurement prior to randomization

   1. For patients < age 18 years: Schwartz formula
   2. For patients ≥ age 18 years: Cockroft-Gault formula
4. Up/c > 1.0 g/g creatinine on first morning void at time of randomization
5. Biopsy confirmed as primary FSGS (including all subtypes) by study pathologist.
6. Steroid resistance: During the last treatment course with high dose steroids prior to randomization, the patient must have demonstrated steroid resistance defined below and not have had a complete remission of proteinuria (Up/c < 0.2 or dipstick urine protein negative/trace) subsequently. The course of steroid treatment that defines resistance must be the same or equivalent to at least 4 weeks of every day dosing with a minimum cumulative dose of 56 mg/kg or 1680 mg of prednisone or its equivalent.
7. May be taking angiotensin-converting enzyme inhibitor (ACEI), angiotensin receptor blocking agent (ARB), vitamin E, or lipid lowering therapy
8. Willingness to comply with clinical trial protocol, medications, and follow-up visits, etc.
9. Screen failure in FSGS-CT based on prior treatment with excluded medication
10. Treatment failure in FSGS-CT based on failure to achieve remission after 26 weeks or 52 weeks of test therapy, i.e., cyclosporine or mycophenolate mofetil (MMF) + oral dexamethasone pulses

Exclusion Criteria

1. Secondary FSGS
2. Treated with cyclophosphamide, chlorambucil, levamisole, methotrexate, nitrogen mustard, or other immunosuppressive medications in the 30 days prior to randomization
3. Lactation, pregnancy, or refusal of birth control in women of child bearing potential
4. Participation in another therapeutic trial concurrently or for 30 days prior to randomization
5. Active/serious infection (including, but not limited to hepatitis B or C, HIV)
6. Malignancy
7. Systemic lupus erythematosus (SLE) or multiple sclerosis
8. Hepatic disease defined as serum AST/ALT > 2.5X the upper limit of normal
9. Patients with blood pressure > 140/95 or > 95th percentile for age/height while receiving maximal doses of 3 or more antihypertensive agents.
10. Diabetes mellitus (DM) type I or II.
11. Hematocrit < 30%
12. Organ transplantation
13. Obesity (based on estimated dry weight at disease onset prior to steroid therapy) defined as:

    1. Body mass index (BMI) > 97th percentile for age if aged 2-20 years
    2. BMI > 40 kg/m2 if aged ≥ 21 years
14. Allergy to study medications
15. Inability to consent/assent

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2005-07; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerance of medications | 16 week treatment period

SECONDARY OUTCOMES:
Reduction in proteinuria | 16 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Howard Trachtman, MD, Principal Investigator — Schneider Children's Hospital of North Shore-LIJ Health System; Debbie Gipson, MD, Principal Investigator — University of North Carolina; Tom Greene, PhD, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Howard Trachtman, New Hyde Park, New York
  - Debbie Gipson, Chapel Hill, North Carolina

REFERENCES:
- [Derived] Liu ID, Willis NS, Craig JC, Hodson EM. Interventions for idiopathic steroid-resistant nephrotic syndrome in children. Cochrane Database Syst Rev. 2025 May 8;5(5):CD003594. doi: 10.1002/14651858.CD003594.pub7. PMID 40337980
- [Derived] Hodson EM, Sinha A, Cooper TE. Interventions for focal segmental glomerulosclerosis in adults. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD003233. doi: 10.1002/14651858.CD003233.pub3. PMID 35224732